CLINICAL TRIAL: NCT00930501
Title: Phase 1 Prospective Study of Markers of Ovarian Reserve in Young Female Cancer Patients
Brief Title: Anti-Mullerian Hormone (AMH) and Antral Follicle Count as Markers of Ovarian Reserve- Prospective Followup of Young Cancer Patients
Acronym: Ovrescancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ariel Revel, MD, Hadassah
Other Study IDs: 111222
Record Dates: First submitted 2009-06-28; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Infertility
Keywords: chemotherapy; cancer; AMH; gonadotoxicity; ovarian reserve; patients exposed to chemotherapy
MeSH Terms: conditions — Infertility; Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bloods
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: women 5-45 yr olf pre and post chemotherapy
  Interventions: Biological: blood tests

INTERVENTIONS:
Biological: blood tests — time 0 is pretreatment time 3, 6 , 9, 12 months from the end of chemotherapy

SUMMARY:
young female cancer patients have improving chances of survival. the main risk is a chronic damage to their ovarian reserve. This may lead to future infertility.

DETAILED DESCRIPTION:
our objective is to prospectively follow patients before and after their cancer treatment. this should help us learn of the gonadotoxicity of various treatments as well as be able to better consult these and future patients of the need of fertility preservation techniques.

ELIGIBILITY:
Inclusion Criteria:

* all females prior and after chemotherapy

Exclusion Criteria:

* do not consent

Ages: 5 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: females 5-45 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Anti mullerian hormone | 2 years

SECONDARY OUTCOMES:
antral follicle count | 2 years
FSH | 2 years
inhibin b | 2 years
menstrual history | 2 years
E2 and prog | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah, Jerusalem, Israel